CLINICAL TRIAL: NCT07150351
Title: The Impact of Anti-Resorptive Agents on Dental Implant Success: An Epidemiological, Meta-Analysis and Retrospective Cohort Study
Brief Title: The Impact of Anti-Resorptive Agents on Dental Implant Success
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202507114RINA
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dental Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study aims to evaluate the relationship between the use of oral anti-resorptive agents and the success rate of dental implants in patients. Medical records from patients who received dental implants between January 2011 and December 2024 at National Taiwan University Hospital were reviewed. The study compares implant success rates between patients who had a history of oral anti-resorptive agents use and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* with complete dental implant records
* patients with or without a history of anti-resorptive agents

Exclusion Criteria:

* patients lacking complete dental radiographic records
* patients in whom the implant site or its relation to the lesion could not be clearly identified

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study population consists of adult patients aged 20 years and older who received dental implant treatment at a single medical center between 2011 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
Dental implant success rate | 12 months after implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan